CLINICAL TRIAL: NCT03430739
Title: Investigating the Optimal Usage Time of Helmet in Babies With Deformational Plagiocephaly
Brief Title: Effect of Usage Time of Helmet in Babies With Deformational Plagiocephaly
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, hhotaman, PhD, Assoc Prof, Trakya University
Other Study IDs: GO 10-76
Record Dates: First submitted 2018-02-06; First posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Non Synostotic Plagiocephaly
Keywords: Deformational Plagiocephaly, Orthotics, Helmet
MeSH Terms: conditions — Plagiocephaly, Nonsynostotic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Babies; Usage time of Helmet between 15-18 hours a day: Babies who worn the helmet for 15-18 hours a day
  Interventions: Other: No intervention
- Babies; Usage time of Helmet between 19-23 hours a day: Babies who worn the helmet for 19-23 hours a day
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Investigating the optimal usage time of helmet therapy is the aim of the study. Participants will be babies with deformational plagiocephaly. Plagiocephalometric assesments will be utilize to follow improvement of head symmetry. Scales asking sensational integration and severity of plagiocephaly will also be used. Time of daily usage will be follow with daily asking the caregivers how long the baby wear the helmet in a day. Participants will follow for three months.

DETAILED DESCRIPTION:
Investigating the optimal usage time of helmet therapy is the aim of the study. Participants will be babies with deformational plagiocephaly. Plagiocephalometric assesments will be utilize to follow improvement of head symmetry. Scales asking sensational integration and severity of plagiocephaly will also be used. Time of daily usage will be follow with daily asking the caregivers how long the baby wear the helmet in a day. Participants will follow for three months. After the follow period completed, participants will be allocated two groups; avarage using 15-18 hours a day and avarage using 19-23 hours a day. Results will be compared for the two groups and correlation between the time of usage and cranial symmetry will be compare.

ELIGIBILITY:
Inclusion Criteria:

have deformational plagiocephaly consent from caregivers age between 1 day to 7 months

Exclusion Criteria:

have another systemic, neurologic or orthopedic problem

Ages: 1 Day to 7 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Babies using helmet due to deformational plagiocephaly.
Sampling Method: Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2018-06-05 (Estimated); Primary Completion 2019-06-05 (Estimated); Study Completion 2019-07-05 (Estimated)

PRIMARY OUTCOMES:
plagiocephaly severity scale | Change from Baseline in head asymmetry at 6th weeks of treatment, at the end of the treatment/12th weeks
  scale which has 5 subgroups as following frontal asymmetry, occipital flattening, head tilt, fascial asymmetry, ear asymmetry

SECONDARY OUTCOMES:
Hemispheric asymmetry | Change from Baseline in head asymmetry at 6th weeks of treatment, at the end of the treatment/12th weeks
  Difference between the right and left hemisphere of head (centimeter)

CONTACTS AND LOCATIONS:
Locations (1):
- Trakya University, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided